CLINICAL TRIAL: NCT01424085
Title: Antibiotic Prophylaxis Before Percutaneous Gastrostomy: A Randomized, Controlled Clinical Trial
Brief Title: Antibiotic Prophylaxis Before Percutaneous Gastrostomy
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Chris Ingraham, Assistant Professor, MD, University of Washington
Other Study IDs: 40912-B
Record Dates: First submitted 2011-08-24; First posted 2011-08-26 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Those receiving antibiotics: Patients who received one prophylactic dose of antibiotics.
- Placebo: Patients who did not receive one prophylactic dose of antibiotics (received placebo).

SUMMARY:
The purpose of this study is to evaluate the use of antibiotics (i.e. Kefzol) before percutaneous gastrostomy performed in interventional radiology. Patient will be randomized to receive antibiotics or placebo before the procedure, and the rates of skin infection after the procedure will be determined between the two groups. This has never been studied in our population of patients undergoing the procedure. However, antibiotics are routinely given despite the lack of evidence. The investigators hypothesize that patient receiving prophylactic antibiotics will have a decreased number of infections compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Anyone over the age of 18 years who is not currently on antibiotics for other reasons

Exclusion Criteria:

* Anyone on antibiotics for the treatment of other infections.
* Anyone under the age of 18 years
* Pregnant patients

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Anyone referred to Interventional Radiology for percutaneous gastrostomy is in the study population (with inclusion and exclusion criteria below).
Sampling Method: Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2012-05; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Rate of infection | Within one month of the procedure (antibiotic dose, if given)
  Wounds surround the g-tube will be assessed at 4 points after the procedure to document the presence of infection. An assessment for redness, induration, pus, etc. will be performed and documented at 4 times points after the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ahmad I, Mouncher A, Abdoolah A, Stenson R, Wright J, Daniels A, Tillett J, Hawthorne AB, Thomas G. Antibiotic prophylaxis for percutaneous endoscopic gastrostomy--a prospective, randomised, double-blind trial. Aliment Pharmacol Ther. 2003 Jul 15;18(2):209-15. doi: 10.1046/j.1365-2036.2003.01684.x. PMID 12869081